CLINICAL TRIAL: NCT02063425
Title: "Evaluation by Transcranial Magnetic Stimulation of the Benefit of Fluoxetine on Motor Recovery After Stroke"
Acronym: EFLUSTIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough recruitment
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D505; 2013-001313-32 (EudraCT Number)
Record Dates: First submitted 2014-01-06; First posted 2014-02-14 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Infarction
Keywords: Motor recovery; Fluoxetine; Transcranial magnetic stimulation; stroke
MeSH Terms: conditions — Cerebral Infarction; Stroke | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine (Active Comparator)
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — 1 pill of 20mg / day, during 3 months
  Other Names: Patients receiving fluoxetine
  Arms: Fluoxetine
Drug: Placebo of fluoxetine — 1 pill of 20mg/day, during 3 months
  Other Names: Patients receiving placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to better characterize the mechanisms of action of fluoxetine in motor recovery and more specifically to identify the neurophysiological substrate underlying fluoxetine-induced motor recovery in stroke.

In this study, the investigators propose to use transcranial magnetic stimulation (TMS) to assess the effect of a chronic treatment of fluoxetine on corticospinal excitability and integrity.

DETAILED DESCRIPTION:
Recently, a phase IIb clinical trial (Chollet et al., 2011 - FLAME study) revealed that early administration of standard-dose oral fluoxetine (a selective serotonin re-uptake inhibitor widely used as antidepressant) to patients with subacute ischaemic stroke and moderate to severe motor deficit in the upper extremity enhanced motor recovery after 3 months, as assessed by the Fugl-Meyer motor scale, suggesting that fluoxetine could be a promising drug to promote recovery in stroke patients. However, the mechanisms, and their specificity, by which fluoxetine improves motor function after stroke remain poorly understood.

The overall objective of this proposal is to better characterize the mechanisms of action of fluoxetine in motor recovery and more specifically to identify the neurophysiological substrate underlying fluoxetine-induced motor recovery in stroke.

The corticospinal system plays a key role in voluntary activation of upper limb muscles. Its integrity has been related to spontaneous (but incomplete) recovery after stroke. So far, the effect of fluoxetine on corticospinal excitability and integrity has been poorly explored although this drug appears promising to promote motor recovery.

In this study, the investigators propose to use transcranial magnetic stimulation (TMS) to assess the effect of a chronic treatment of fluoxetine on corticospinal excitability and integrity. The investigators believe that this approach will be suitable to determine the mechanisms of action of this drug on motor recovery after stroke.

The investigators will assess in a double-blind, monocentric (Saint-Anne Hospital Stroke center), randomised, placebo-controlled study, the effect of a chronic treatment of fluoxetine on corticospinal excitability and integrity using TMS in 40 patients suffering from ischaemic stroke with hemiplegia or hemiparesis affecting motor hand functions.

By coupling TMS, visuomotor grip tracking task and several clinical scales, the investigators' results will allow a more system-specific assessment than the Fugl-Meyer motor scale of fluoxetine-induced motor hand recovery in stroke. We believe that this study will support the beneficial effect of fluoxetine to promote motor recovery in stroke and will open new vistas for treatment options using fluoxetine in patients with motor impairments. It is expected that this study will provide preliminary data that will be subsequently used to design new, more focused, clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Man and women, aged from 18 to 80 years.
* Social security affiliation
* Inclusion from day 3 to day 15 after stroke or brain haemorrhage
* Hemiparesia with upper limb motor deficit (Fugl-Meyer score - hand < or = 10)
* Informed consent

Exclusion Criteria:

* Score NIHSS > 20
* Depression (criteria DSM5-R) with MADRS score > 19
* History of recurrent bipolar or depressive disorders.
* History of behavior or suicidal idea
* Family history of extension of the interval QT or congenital long interval QT
* History of clinical stroke
* Aphasia preventing correct evaluation of motor and depression scales.
* Patients treated by antidepressant drugs, monoamine oxidase inhibitor (IMAO), and neuroleptics in the past month
* Benzodiazepines within 48 hours preceding inclusion.
* Intolerance or allergy to fluoxetine (Sandoz® 20 mg pill)
* Severe swallowing disorders preventing oral administration of the treatment
* Planned carotid surgery
* Pregnant or breast-feeding woman
* Hepatic failure (TGO and TGP >2N); severe renal failure (creatinine >180micromol/l)
* Concomitant severe disease not allowing follow-up.
* Participation to another therapeutic study.
* Contraindication to MRI and TMS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Slope of the curve of recruitment of the PEMs | M3
  Significant difference, between the treated group and the group control, of the slope of the curve of recruitment of the PEMs between the beginning (D0) and the end of the treatment (processing) (M3).

SECONDARY OUTCOMES:
Slope of recruitment of the PEMs | D0, M3, M6
  Effect of a first dose of fluoxétine on the slope of recruitment of the PEMs.
Slope of recruitment of the PEMs | D0, M3, M6
  Persistence of fluoxétine effect on the slope of recruitment of the PEMs to M6.
Index finger force control in paretic hand under time-course of treatment of Fluoxetine | D0, M3, M6
  A visuomotor tracking task is used to measure accuracy of force control (NewtonSecond, Ns) and time taken to release force (release duration, ms). Performance between time-points will be measured (Ns, before-after treatment).
  Effects of fluoxetine on force control parameters (e.g., accuracy and release duration) in paretic hand.
in index finger force control in non-paretic hand under time-course of treatment of Fluoxetine | D0, M3, M6
  Same visuomotor tracking mesures as above but acquired in non-paretic hand. Effects of fluoxetine on the non-affected hand (error, Ns; release duration, ms).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BARON, MD, Study Director — Centre Hospitalier Sainte-Anne
Locations (1):
- Centre Hospitalier Sainte-Anne, Paris, France